CLINICAL TRIAL: NCT00430794
Title: A Randomised, Placebo Controlled Trial of the Efficacy of the Addition of Spironolactone to Modern Antihypertensive Treatment Regimens in Patients With Resistant Hypertension
Brief Title: The Efficacy of Spironolactone in Patients With Resistant Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties with recruitment.
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH14399
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2010-12-06 (Estimated); Status verified 2007-02

CONDITIONS: Hypertension
Keywords: resistant hypertension; Spironolactone; double-blind; randomised controlled trial; ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension | interventions — Spironolactone

INTERVENTIONS:
Drug: Spironolactone

SUMMARY:
To determine the efficacy of the addition of spironolactone to modern blood pressure lowering treatment regimens in patients with resistant hypertension (whose blood pressure is uncontrolled despite three blood pressure lowering drugs)

DETAILED DESCRIPTION:
Objective: To assess the antihypertensive efficacy of adding spironolactone to the antihypertensive treatment of patients with resistant hypertension.

Background and Rationale: The proportion of hypertensive patients meeting the definition of resistant hypertension is growing rapidly as doctors use more combination antihypertensive treatments in order to reach lower target blood pressures. Spironolactone is often used in specialist clinics for patients with resistant hypertension although it is currently only licensed in the UK for use in hypertension complicated by primary hyperaldosteronism. Uncontrolled studies suggest that spironolactone is a very effective antihypertensive in the modern management of resistant hypertension but we could find no randomised trials in this setting. In the Sheffield Hypertension Clinic spironolactone is currently used as one of the drugs of choice in patients with resistant hypertension, particularly in women and is anecdotally often very effective.

Study methods. The study will be a double- blind randomised placebo controlled trial with a parallel group design assessing the addition of 25mg spironolactone to existing antihypertensive treatment, titrated to 50mg if necessary in 40 patients with resistant hypertension (20 patients per group) over a period of 6 weeks. Resistant hypertension will be defined as: blood pressures not adequately controlled (systolic blood pressure (SBP) >140 mmHg and/or diastolic blood pressure (DBP) >85 mmHg in clinic and on ambulatory blood pressure monitoring) despite treatment with the maximum tolerated dose of three antihypertensive agents. All patients' current antihypertensive treatment will include a thiazide diuretic and at least one of a beta-blocker, angiotensin converting enzyme inhibitor or angiotensin II receptor antagonist. The primary endpoint will be the difference between the spironolactone and placebo groups in change in daytime average systolic blood pressure on 24-hour ambulatory blood pressure monitoring from day 0 to day 42.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Hypertension (essential or secondary) managed in Sheffield Hypertension Clinic or general practice or both.
* Blood pressures not adequately controlled (systolic blood pressure (SBP) >140 mmHg and/or diastolic blood pressure (DBP) >85 mmHg in clinic and on ambulatory blood pressure monitoring) despite treatment with the maximum tolerated dose of three antihypertensive agents.
* Additional antihypertensive treatment deemed appropriate by the patients' doctor.
* Patients' current antihypertensive treatment includes a thiazide diuretic and at least one of a beta-blocker, angiotensin converting enzyme inhibitor or angiotensin II receptor antagonist.

Exclusion Criteria:

* Definite indication or contraindication for spironolactone
* Known Conn's syndrome (definite indication for spironolactone)
* Heart failure NYHA class III or IV (definite indication for spironolactone)
* Known hepatic failure or significant cirrhosis
* Known pregnancy or women planning pregnancy
* Women of child bearing potential not using adequate contraceptive methods
* Serum creatinine > 221µmol/l
* Serum Potassium > 5.0mmol/l
* Clinic blood pressure or daytime ambulatory blood pressure >240/120

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-03; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the difference between the spironolactone and placebo groups in change in daytime average systolic blood pressure on ABPM from day 0 to day 42

SECONDARY OUTCOMES:
Difference between the spironolactone and placebo groups in change in daytime average diastolic blood pressure on ABPM from day 0 to day 42
Difference between the spironolactone and placebo groups in change in systolic and diastolic clinic blood pressure (mean of 2nd and 3rd readings) from day 0 to day 42
Difference between the spironolactone and placebo groups in change in serum creatinine from day 0 to day 42
Difference between the spironolactone and placebo groups in change in serum potassium from day 0 to day 42
Difference between the spironolactone and placebo groups in change in body weight from day 0 to day 42

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Jackson, MB ChB, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Clinical Research Facility, Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom